CLINICAL TRIAL: NCT03700138
Title: Prospective, Randomised, Placebo-controlled Study of Polyvalent Intravenous Immunoglobulins for the Treatment of Primary Sjögren's Syndrome Associated Painful Sensory Neuropathies
Brief Title: Intravenous Immunoglobulins for the Treatment of Primary Sjögren's Syndrome Associated Painful Sensory Neuropathies
Acronym: TINISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6621
Record Dates: First submitted 2018-08-24; First posted 2018-10-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Primary Sjögren's Syndrome Painful Sensory Neuropathies
MeSH Terms: interventions — Immunoglobulins, Intravenous; Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Privigen (Experimental): TThe treatment (IV Ig, 100mg/ml at the dose of 2g/kg of body weight) will be administered by perfusion every 6 weeks, with a total of 3 perfusions administered (W0, W4, W8).
  Interventions: Drug: Privigen® 100mg/ml at the dose of 2g/kg of body weight
- Placebo (Placebo Comparator): The treatment (NaCl 0,9% 20 ml/kg) will be administered by perfusion every 4 weeks, with a total of 3 perfusions administered (W0, W4, W8).
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: Privigen® 100mg/ml at the dose of 2g/kg of body weight — The treatment (IV Ig, 100mg/ml at the dose of 2g/kg of body weight) will be administered by perfusion every 4 weeks, with a total of 3 perfusions administered (W0, W4, W8).
  Arms: Privigen
Drug: NaCl 0,9% — The treatment (NaCl 0,9% 20 ml/kg) will be administered by perfusion every 4 weeks, with a total of 3 perfusions administered (W0, W4, W8).
  Arms: Placebo

SUMMARY:
To summarise, the peripheral neurological complications experienced by patients with primary Sjögren's syndrome are particularly bothersome since they are common and often result in significant disability related to pain or motor impairment. There is currently no standard treatment for these patients.

As these neuropathies are caused by an immune system dysfunction, which is related to a variety of different pathogenic mechanisms, the use of immunosuppressant or immunomodulator drugs is often justified.

With the exception of the vascularitis-related multiplex mononeuropathies, other pSS-related neuropathies could be suitable candidates for IV Ig treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 80 years
* Primary Sjögren's syndrome defined as per the European and American criteria (5)
* Peripheral neuropathy clinically defined:

  * Pure sensitive (lymph node disease) or sensorimotor neuropathies
  * Proved EMG
* Renal function, and viral evaluation (VIH and hepatitis serology) :

  *Clairance > 50 (In case of biological abnormality, the second dosage can be scheduled within 2 weeks)
* Effective contraception during the study period
* Patient capable of understanding information about the study and of giving his/her consent
* Patient informed of the preliminary medical exam results
* Patient with healthcare insurance
* Written consent signed

Exclusion Criteria:

* Peripheral neurological damage of the type vascularitis-related multiplex mononeuropathy
* Small fibers neuropathy
* Neuropathy suspected of being related to alcohol, diabetes or post-chemotherapy
* Chronic viral infection (HCV, HBV, HIV, etc.)
* Prior treatment with polyvalent intravenous immunoglobulins in the 6 months preceding the study
* Corticosteroid treatment at a dose greater than 20 mg/d of prednisone equivalent or no stable dose for at least 1 month before inclusion
* Conventional immunosuppressant treatment with azathioprin, cyclophosphamide or mycophenolate mofetil on-going or interrupted less than one month before inclusion
* Rituximab or other biotherapy (belimumab, tocilizumab, …) less than 6 months before the start of the study treatment
* Immunomodulating treatment with methotrexate no stable dose for at least 2 months before inclusion
* Hydroxychloroquine no stable dose for at least 3 months before inclusion
* Pilocarpine hydrochloride secretagogue treatment no stable dose for at least one month before inclusion
* Treatment with amitriptyline, clomipramine, carbamazepine, clonazepam, pregabaline, duloxetine or gabapentine if the dose has not been stable for at least one month before inclusion (possible dose reduction to be documented).
* renal clairance < 50 ml/mn
* HIV seropositivity
* HBV, or HCV viral replication
* Contraindication to the use of IV Ig: h Hypersensitivity to the active substance or to any of the excipients; hypersensitivity to human immunoglobulins, especially in patients with antibodies against IgA; patients with hyperprolinaemia.
* Contraindication to the use of Nacl
* Immunization with live attenuated vaccine within 2 weeks prior to inclusion
* Participation in a clinical study with an investigational product with an exclusion period
* Women of child bearing potential or intends to become pregnant, unless they are using an effective method of birth control* and a βHCG blood test negative
* Pregnant or nursing (lactating) women
* Patient under legal guardianship
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Improvement of at least 20% over placebo of numerical Pain Scale | At week 11
Improvement of at least 20% over placebo with the R-DS scale (Rasch-built Overall Disability Scale) | At week 11

SECONDARY OUTCOMES:
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. | Weeks 11
  o Quality of life scale (SF 36)
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. | Weeks 11
  o HAD depression score
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. | Weeks 11
  o Numerical Fatigue Scale
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. | Weeks 11
  o A fatigue scale (EMIF)
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. intensity. | Weeks 11
  o Numerical Dry mouth Scale
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. intensity. | Weeks11
  o Numerical Dry eye Scale
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. | Weeks 11
  o ESSPRI
Evaluate patient's quality of life, fatigue, and Sicca syndrome intensity. | Weeks 11
  o ESSDAI
Evaluate intensity of the IV Ig effect on neurological scales | Weeks 11
  o Overall Neuropathy Limitations Scale (ONLS)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques-Eric Jacques-Eric, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France